CLINICAL TRIAL: NCT04930549
Title: Impact of Dapagliflozin on Vascular Function in Chronic Kidney Disease Patients
Brief Title: Vascular Impact of Dapagliflozin in CKD Patients (DAPAVASC)
Acronym: DAPAVASC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021/0188/HP
Record Dates: First submitted 2021-06-03; First posted 2021-06-18 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2022-11

CONDITIONS: Renal Insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin 10Mg Tab (Experimental): Dapagliflozin 10 mg film-coated tablets
  Interventions: Drug: Dapagliflozin 10Mg Tab; Procedure: impedance cardiography; Procedure: Applanation tonometry; Procedure: post-ischemic hyperemia of forearm; Procedure: haemodynamics parameters
- Placebo (Placebo Comparator): Identical film-coated tablets without dapagliflozin
  Interventions: Drug: Placebo; Procedure: impedance cardiography; Procedure: Applanation tonometry; Procedure: post-ischemic hyperemia of forearm; Procedure: haemodynamics parameters

INTERVENTIONS:
Drug: Dapagliflozin 10Mg Tab — Patients receive dapagliflozin 10mg tablets once a day during 12 weeks
  Arms: Dapagliflozin 10Mg Tab
Drug: Placebo — Patients receive placebo tablets once a day during 12 weeks
  Arms: Placebo
Procedure: impedance cardiography — impedance cardiography (PhysioFlow® PF-05 Lab1TM, Manatec Biomedical) is done for evaluation of cardiac function
Procedure: Applanation tonometry — Applanation tonometry will be done using SphygmoCor®, Hogimed) is done for evaluation of arterial stiffness
Procedure: post-ischemic hyperemia of forearm — An arterial occlusion cuff will be placed on the forearm, and will be deflated to allow post-ischemic hyperemia with the continuous measurements of brachial artery diameter and blood flow velocity by high-resolution echotracking coupled to a Doppler system (ArtLab system®)
Procedure: haemodynamics parameters — haemodynamics parameters will be evaluated using automatic oscillometric recorder

SUMMARY:
This study aims to determine whether dapaglfiflozin 12-week administration is associated with a beneficial impact on the vasculature of patients with chronic kidney disease.

DETAILED DESCRIPTION:
A prospective, randomized, double-blind studies evaluating the impact of once-daily dapagliflozin 10 mg versus placebo for 12 weeks on endothelial function, as primary endpoint, will be conducted in 56 patients with chronic kidney disease (eGFR ≥25 and ≤60 mL/min/1.73m2 by CKD-EPI) and without diabetes (fasting glycemia≥1.26 mg/dL, oral hypoglycemic agents or insulin) on top of standard treatment (n=27 per group). Indexes of arterial stiffness, cardiovascular coupling, cardiac function and plasma concentrations of endothelial, inflammatory and oxidative stress biomarkers will be assessed as secondary endpoints. Patients will be recruited in the Departments of Cardiology and Nephrology of Rouen University Hospital. The study will include an inclusion visit (V1), 2 exploration visits performed before (V2) and 12 weeks (V3) after treatment initiation, and 1 output study (V4).

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease (eGFR ≥25 and ≤60 mL/min/1.73m² by CKD-EPI)
* Age ≥ 18 years
* Receiving a stable dose of an ACE inhibitor or ARB for at least 12 weeks before screening or patients who were documented to be intolerant to ACE inhibitors or ARBs

Exclusion Criteria:

* Type 1 and type 2 diabetes (fasting glycemia≥126 mg/dL or use of oral hypoglycemic agents or insulin)
* Recessive or autosomal dominant polycystic kidney disease
* Anti-neutrophil cytoplasmic antibody (ANCA)-associated vasculitis
* Lupus nephritis
* Receiving cytotoxic therapy, immunosuppressive therapy or other immunotherapy for primary or secondary renal disease within 6 months prior to enrolment
* History of organ transplantation
* Body weight > 35 kg/m²
* Receiving therapy with a sodium glucose co-transporter 2 (SGLT2) inhibitor within 8 weeks prior to enrolment or previous intolerance of an SGLT2 inhibitor
* Patients with NYHA class IV congestive heart failure at the time of enrolment
* Myocardial infarction, unstable angina, stroke or transient ischemic attack (TIA) within 12 weeks prior to enrolment
* Coronary revascularization (percutaneous coronary intervention or coronary artery bypass grafting) or valvular repair/replacement within 12 weeks prior to enrolment or is planned to undergo any of these procedures after randomization
* Active malignancy requiring treatment at the time of enrolment or is planned to undergo any treatment after randomization
* Severe hepatic impairment (Child-Pugh class C)
* History of frequent genital mycotic infections (>2)
* Current pregnancy OR women of child-bearing potential (ie, those who are not chemically or surgically sterilized or who are not post-menopausal) who are not willing to use a medically accepted method of contraception that is considered reliable in the judgment of the investigator OR women who have a positive pregnancy test at enrolment or exploration visits OR women who are breast-feeding
* Contraindications to use glyceryl trinitrate (in particular allergy to nitrates or concomitant use of vasodilators)
* Participation in another clinical study with an investigational product during the last month prior to enrolment
* Inability of the patient, in the opinion of the investigator, to understand and/or comply with procedures and/or follow-up OR any conditions that, in the opinion of the investigator, may render the patient unable to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline of brachial artery endothelial function using echography | 12 weeks
  Change in brachial artery flow-mediated dilatation in response to post-ischemia hyperemia using difference of brachial artery diameter

SECONDARY OUTCOMES:
Change from baseline of arterial stiffness using applanation tonometry | 12 weeks
  Change in carotid-to-femoral pulse wave velocity
Change from baseline of carotid artery geometry using echography (1) | 12 weeks
  Change in carotid diastolic diameter
Change from baseline of carotid artery geometry using echography (2) | 12 weeks
  Change in carotid intima-media thickness using echography
Change from baseline of cardiac function by impedance cardiography (1) | 12 weeks
  Change in cardiac output
Change from baseline of cardiac function by impedance cardiography (2) | 12 weeks
  Change in stroke volume
Change from baseline of cardiac function by impedance cardiography (3) | 12 weeks
  Change in ejection fraction
Change from baseline of cardiac function by impedance cardiography (4) | 12 weeks
  Change in end-diastolic volume
Change from baseline of cardiac function by impedance cardiography (5) | 12 weeks
  Change in total peripheral resistance,
Change from baseline of cardiac function by impedance cardiography (6) | 12 weeks
  Change in left ventricular end-systolic elastance
Change from baseline of epoxyeicosatrienoic acid bioavailability | 12 weeks
  Change in epoxyeicosatroenoic acid bioavailibility during heating
Change from baseline of plasma NO bioavailability | 12 weeks
  Change in plasma nitrite bioavailibility during heating

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Guerrot, MD, PhD, Principal Investigator — University Hospital, Rouen; Jeremy Bellien, PharmD, PhD, Study Director — University Hospital, Rouen
Locations (2):
- France (2):
  - Department of Nephrology, Bois-Guillaume
  - Department of Pharmacology, Rouen

IPD SHARING:
Plan to Share IPD: No